CLINICAL TRIAL: NCT05303298
Title: Evaluating Gastro-oesophageal Reflux After Palliative Stenting for Malignant Distal Oesophageal Obstruction Using Anti-Reflux Stents: a Randomised Controlled Trial
Brief Title: Evaluating Acid Reflux After Oesophageal Stenting Using Anti-reflux Stents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Matthias Scriba, Senior Registrar: Upper Gastrointestinal Surgery, Surgical Gastroenterology, Department of Surgery, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HREC REF NO: 706/2021
Record Dates: First submitted 2022-02-28; First posted 2022-03-31 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Cancer; Reflux, Gastroesophageal
Keywords: Esophageal Cancer; Palliative Stenting; Gastroesophageal Reflux; Anti-reflux Stents
MeSH Terms: conditions — Esophageal Neoplasms; Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to receive either an anti-reflux oesophageal stent or a conventional oesophageal stent.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will remain unaware of which type of stent they have received. Follow-up will be performed telephonically and the Outcomes Assessor will also remain blinded as to what type of stent the participant received
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anti-reflux Oesophageal Stent Group (AOSG) (Experimental): All patients randomised to this arm will receive an anti-reflux fully covered self-expanding metal oesophageal stent
  Interventions: Device: Anti-reflux oesophageal stent
- Conventional Oesophageal Stent Group (COSG) (Active Comparator): All patients randomised to this arm will receive a conventional fully covered self-expanding metal oesophageal stent that does not contain an anti-reflux mechanism
  Interventions: Device: Conventional oesophageal stent

INTERVENTIONS:
Device: Anti-reflux oesophageal stent — Fully covered self-expanding metal stent with anti-reflux mechanism
  Arms: Anti-reflux Oesophageal Stent Group (AOSG)
Device: Conventional oesophageal stent — Fully covered self-expanding metal stent without an anti-reflux mechanism
  Arms: Conventional Oesophageal Stent Group (COSG)

SUMMARY:
Incurable oesophageal cancer remains a global problem and in South Africa the vast majority of patients with oesophageal cancer have advanced disease at first presentation and are not curable. Likely the most distressing symptom of advanced cancer in the oesophagus is dysphagia, which is the inability to swallow solids and later also liquids. This is successfully addressed in most cases by the placement of a stent in the oesophagus which opens the area of obstruction. When placed in the lower oesophagus, one of the major drawbacks of these stents is that they disrupt the anti-reflux mechanism of the oesophago-gastric junction, which can result in severe acid reflux, severely impacting the quality of life of the patient. To address this problem, a range of approved anti-reflux stents have been developed and tested in numerous trials. To date, the evidence is conflicting and there is insufficient current evidence to support the routine use of these stents. However, the trials are not all similar in how the acid reflux was measured or what type of stent was used. Furthermore, the use of anti-reflux medication, such as proton pump inhibitors, which may help reduce reflux, are not standardised across the trials and make further conclusions about these stents difficult to interpret.

No data from Sub-Saharan Africa on the use of anti-reflux stents in these patients is available. South Africa faces a large burden of incurable oesophageal cancer and improving the quality of life of these patients is of paramount importance. This randomised controlled trial aims to investigate whether anti-reflux stents do indeed reduce acid reflux in patients with incurable oesophageal cancer compared to conventional oesophageal stents that do not have such an anti-reflux mechanism. Reflux will be measured using patient questionnaires about reflux, and other quality of life parameters, and will also be objectively measured using oesophageal scintigraphy, which has not been used in previous similar trials.

DETAILED DESCRIPTION:
Oesophageal cancer is an aggressive condition, resulting in the vast majority of patients having evidence of locally invasive, irresectable disease or distant metastases at the time of presentation. Overall survival remains poor. Management in the South African setting is plagued by late presentation of these patients, with less than 5% being eligible for curative treatment and median survival from the time of diagnosis being only 15 weeks, while those who present with complete obstruction having a median survival of only 75 days (10.7 weeks). Treatment of these patients in the South African setting remains predominantly palliative. The most common and debilitating symptom of advanced oesophageal malignancy is progressive dysphagia, which can be addressed by the endoscopic placement of self-expanding metal stents. The major drawback of stenting tumours in the lower oesophagus or oesophagogastric junction (OGJ), is the associated gastro-oesophageal reflux (GOR) resulting from the stent crossing the lower oesophageal sphincter and essentially negating the native anti-reflux mechanism. Significant reflux is the most common complaint worsening quality of life after stent placement in these patients and can be as high as 100% in some series. Prescribing routine proton pump inhibitors (PPIs) or placing stents with built-in anti-reflux mechanisms are methods aimed at reducing this symptomatic reflux.

Theoretically, oesophageal stents containing an anti-reflux valve should provide a physical barrier to prevent gastric content (which may be acidic or non-acidic) refluxing into the oesophagus, but whether this results in decreased rates of GOR in reality is somewhat controversial. To date, a number of trials have compared a range of anti-reflux oesophageal stents to conventional oesophageal stents and although there have been some conflicting results, a systematic review and meta-analysis in 2019 concludes that GOR is not significantly reduced by the use of anti-reflux stents. However, there are a number of factors that must be mentioned before this conclusion can be applied to dictate clinical practice. Firstly, the included trials all have reasonably small participant numbers, with 65 patients being the highest number of patients enrolled in any of these trials. In fact, the authors conclude that the meta-analysis is underpowered. Furthermore, the type of anti-reflux stent used varies with almost every trial and may well influence efficacy of reducing GOR. Anti-reflux medical therapy such as the use of proton pump inhibitors (PPIs) also varied greatly amongst the studies. Some prescribed PPIs only to the conventional stent group, others did not use PPIs in either group, while the rest did not mention whether PPIs were routinely given or not. This could possibly influence symptomatic reflux and act as a significant confounding factor.

The measurement of GOR in the trials assessed in this meta-analysis shows significant heterogeneity, with some studies using patient questionnaires (some of these assess quality of life in general and do not specifically focus on reflux symptoms), others use contrast oesophagography or functional 24-hour pH monitoring. These additional factors make the results of this underpowered meta-analysis difficult to interpret. Since then, a further randomised controlled trial (RCT) was conducted by Dua et al. This included a total of 60 patients, comparing a novel tricuspid-shaped valve anti-reflux stent (30 patients) to conventional stenting (30 patients). Importantly, this trial was a non-inferiority trial to assess safety and efficacy at improving dysphagia for the new stent. Assessment of GOR was a secondary outcome and although reflux rates favoured the new anti-reflux stent, this did not reach statistical significance. The current level I and II evidence on reducing GOR with anti-reflux stents is thus not definitive and leaves the topic unresolved.

While research in high income countries is focused on the management of early oesophageal malignancies, this is not appropriate in the South African setting where the vast majority of patients are irresectable at initial presentation. Local research is significantly limited and there is a paucity of data from South Africa, and Africa as a whole, as regards the palliative management of malignant oesophageal dysphagia. Specific evidence on the use of anti-reflux stents is absent. Further research is thus invaluable in assessing if the palliative care of these patients can be improved by using anti-reflux stents.

This prospective randomised controlled trial aims to compare the incidence of symptomatic volume GOR after the use of anti-reflux oesophageal covered metal stents versus conventional oesophageal covered metal stents for lower oesophageal malignant strictures in a South African tertiary referral centre with a high rate of palliative stenting for advanced oesophageal carcinoma. Reflux will be assessed subjectively by the administration of patient questionnaires aimed at identifying severity of acid reflux, but also the degree of dysphagia, pain and coughing before and after stent placement. Reflux will also be assessed objectively by using oesophageal scintigraphy performed shortly after stent insertion. Scintigraphy has not previously been used to measure GOR in these patients and is chosen for its accuracy and non-invasive nature (compared to, for example, pH monitoring which requires the placement of an uncomfortable nasal probe for 24 hours and is considered inappropriate in this cohort where the main focus lies on quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients - 18 years of age or older
* Informed consent obtained from the patient after oral and written explanation of the trial
* Histologically confirmed malignancy of the distal oesophagus or OGJ
* Obstructive or irresectable malignancy due to metastases, local tumour infiltration or poor performance status
* Once deployed, the distal end of the stent must have crossed the OGJ junction and be lying within the proximal stomach

Exclusion Criteria:

* Patient declining or unable to give informed consent, including inability to speak or understand either English, Afrikaans or isiXhosa (the three most commonly spoken local languages).
* Patient unable to comply with the follow-up protocol of the trial (e.g. does not have a contactable telephone number)
* Oesophageal cancers selected for curative treatment or irresectable oesophageal cancers selected for palliative chemoradiation, but not requiring oesophageal stenting
* Benign oesophageal pathology or extrinsic compression of the oesophagus from another cause
* Patients with oesophageal cancers where the stent does not cross the OGJ
* Pregnant patients
* Patient performance status precluding any intervention or sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Subjective gastro-oesophageal reflux (GOR) - change in GOR over specified time periods | Will be assessed pre-intervention and then at 1, 2, 4, and 8 weeks post intervention
  Self-reported symptomatic reflux using a validated reflux patient questionnaire - the GerdQ questionnaire. GerdQ: score ranges from 0 - 18 points with higher scores equating to higher GOR rates.
Objective gastro-oesophageal reflux (GOR) | Will be performed as a once-off investigation on day 1 post stenting
  Objective measure of GOR will be done using oesophageal scintigraphy

SECONDARY OUTCOMES:
Dysphagia - change in dysphagia over specified time periods | Will be assessed pre-intervention and then at 1, 2, 4, and 8 weeks post intervention
  Dysphagia will be assessed pre- and post intervention using a validated 5 part dysphagia score described by Knyrim et al - scores are reported as 0 - 5, with higher scores indicating more severe dysphagia.
Pain - Change in pain over specified time periods | Will be assessed pre-intervention and then at 1, 2, 4, and 8 weeks post intervention
  Pain will be assessed using a validated visual analog pain score using pictures of faces to signify pain. Pain will be rated from 0 - 5, with higher scores indicating more severe pain
Cough - change in pain over specified time periods | Will be assessed pre-intervention and then at 1, 2, 4, and 8 weeks post intervention
  Cough will be assessed using a validated cough score, the Simplified Cough Score assessing both daytime and night-time cough severity. Score will range from 0 - 6, with higher score indicating worse cough symptoms.
Stent-related complications | Documentation will occur at the time of stent insertion, day 1 post insertion and then at scheduled follow-ups at weeks 1, 2, 4 and 8 post-insertion or aat any time during the study period if a stent-related complication is reported
  All complications related to the stent insertion and later complications related to the stent will be documented
Survival | Documented at 8 weeks post stent insertion
  Participant survival will be documented at the end of the study period

CONTACTS AND LOCATIONS:
Overall Officials: Matthias F Scriba, FCS (SA), Principal Investigator — University of Cape Town
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) that underlie the results reported in the published article for this study, after deidentification, will be made available to any investigator or investigators who request the data for analyses to achieve specific aims of a proposed research study. The study and proposed use of the data must be approved by an independent review committee identified for this purpose. The Study Protocol and Informed Consent Form will also be made available on request. Data will be available immediately after publication of the study and for 5 years after this. Proposals should be directed to matthias.scriba@gmail.com. to gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available immediately after publication of the study and for 5 years after this.
Access Criteria: The study and proposed use of the data must be approved by an independent review committee identified for this purpose. Proposals should be directed to matthias.scriba@gmail.com. to gain access, data requestors will need to sign a data access agreement. Requests will be assessed by the study's Primary Investigator (PI) and the Study Sponsor, the University of Cape Town.

REFERENCES:
- [Background] Pandit S, Samant H, Morris J, Alexander SJ. Efficacy and safety of standard and anti-reflux self-expanding metal stent: A systematic review and meta-analysis of randomized controlled trials. World J Gastrointest Endosc. 2019 Apr 16;11(4):271-280. doi: 10.4253/wjge.v11.i4.271. PMID 31040888
- [Background] Ferndale L, Sartorius B, Aldous C, Thomson SR. Oesophageal cancer in Area 2 of Kwazulu-Natal: predictors of late presentation. S Afr J Surg. 2019 Jun;57(2):4-9. PMID 31342677
- [Background] Nel D, Omar M, Chinnery G, Jonas E. Disparity in oesophageal cancer management in South Africa: a comparison between two tertiary centres with special focus on the palliation of dysphagia. S Afr J Surg. 2019 Jun;57(2):10-15. PMID 31342678
- [Background] Ferndale L, Aldous C, Hift R, Thomson S. Gender Differences in Oesophageal Squamous Cell Carcinoma in a South African Tertiary Hospital. Int J Environ Res Public Health. 2020 Sep 28;17(19):7086. doi: 10.3390/ijerph17197086. PMID 32998198
- [Background] Dandara C, Robertson B, Dzobo K, Moodley L, Parker MI. Patient and tumour characteristics as prognostic markers for oesophageal cancer: a retrospective analysis of a cohort of patients at Groote Schuur Hospital. Eur J Cardiothorac Surg. 2016 Feb;49(2):629-34. doi: 10.1093/ejcts/ezv135. Epub 2015 Apr 12. PMID 25870217
- [Background] Dua KS, DeWitt JM, Kessler WR, Diehl DL, Draganov PV, Wagh MS, Kahaleh M, Wong Kee Song LM, Khara HS, Khan AH, Aburajab MM, Ballard D, Forsmark CE, Edmundowicz SA, Brauer BC, Tyberg A, Buttar NS, Adler DG. A phase III, multicenter, prospective, single-blinded, noninferiority, randomized controlled trial on the performance of a novel esophageal stent with an antireflux valve (with video). Gastrointest Endosc. 2019 Jul;90(1):64-74.e3. doi: 10.1016/j.gie.2019.01.013. Epub 2019 Jan 23. PMID 30684601
- [Background] Jones R, Junghard O, Dent J, Vakil N, Halling K, Wernersson B, Lind T. Development of the GerdQ, a tool for the diagnosis and management of gastro-oesophageal reflux disease in primary care. Aliment Pharmacol Ther. 2009 Nov 15;30(10):1030-8. doi: 10.1111/j.1365-2036.2009.04142.x. Epub 2009 Sep 8. PMID 19737151
- [Background] Blomberg J, Wenger U, Lagergren J, Arnelo U, Agustsson T, Johnsson E, Toth E, Lagergren P. Antireflux stent versus conventional stent in the palliation of distal esophageal cancer. A randomized, multicenter clinical trial. Scand J Gastroenterol. 2010;45(2):208-16. doi: 10.3109/00365520903443860. PMID 19968614
- [Background] Coron E, David G, Lecleire S, Jacques J, Le Sidaner A, Barrioz T, Coumaros D, Volteau C, Vedrenne B, Bichard P, Boustiere C, Touchefeu Y, Bregeon J, Prat F, Le Rhun M; Societe Francaise d'Endoscopie Digestive (SFED). Antireflux versus conventional self-expanding metallic Stents (SEMS) for distal esophageal cancer: results of a multicenter randomized trial. Endosc Int Open. 2016 Jun;4(6):E730-6. doi: 10.1055/s-0042-106960. PMID 27556085
- [Background] Shim CS, Jung IS, Cheon YK, Ryu CB, Hong SJ, Kim JO, Cho JY, Lee JS, Lee MS, Kim BS. Management of malignant stricture of the esophagogastric junction with a newly designed self-expanding metal stent with an antireflux mechanism. Endoscopy. 2005 Apr;37(4):335-9. doi: 10.1055/s-2005-861113. PMID 15824943
- [Background] Sabharwal T, Gulati MS, Fotiadis N, Dourado R, Botha A, Mason R, Adam A. Randomised comparison of the FerX Ella antireflux stent and the ultraflex stent: proton pump inhibitor combination for prevention of post-stent reflux in patients with esophageal carcinoma involving the esophago-gastric junction. J Gastroenterol Hepatol. 2008 May;23(5):723-8. doi: 10.1111/j.1440-1746.2008.05396.x. PMID 18410607
- [Background] Power C, Byrne PJ, Lim K, Ravi N, Moore J, Fitzgerald T, Keeling PW, Reynolds JV. Superiority of anti-reflux stent compared with conventional stents in the palliative management of patients with cancer of the lower esophagus and esophago-gastric junction: results of a randomized clinical trial. Dis Esophagus. 2007;20(6):466-70. doi: 10.1111/j.1442-2050.2007.00696.x. PMID 17958720
- [Background] Homs MY, Wahab PJ, Kuipers EJ, Steyerberg EW, Grool TA, Haringsma J, Siersema PD. Esophageal stents with antireflux valve for tumors of the distal esophagus and gastric cardia: a randomized trial. Gastrointest Endosc. 2004 Nov;60(5):695-702. doi: 10.1016/s0016-5107(04)02047-4. PMID 15557944
- [Background] Blum D, Selman LE, Agupio G, Mashao T, Mmoledi K, Moll T, Dinat N, Gwyther L, Sebuyira LM, Ikin B, Downing J, Kaasa S, Higginson IJ, Harding R. Self-report measurement of pain & symptoms in palliative care patients: a comparison of verbal, visual and hand scoring methods in Sub-Saharan Africa. Health Qual Life Outcomes. 2014 Aug 2;12:118. doi: 10.1186/s12955-014-0118-z. PMID 25085579
- [Background] Lai K. Chinese National Guidelines on Diagnosis and Management of Cough: consensus and controversy. J Thorac Dis. 2014 Oct;6(Suppl 7):S683-8. doi: 10.3978/j.issn.2072-1439.2014.10.06. No abstract available. PMID 25383201
- [Background] Maurer AH, Parkman HP. Update on gastrointestinal scintigraphy. Semin Nucl Med. 2006 Apr;36(2):110-8. doi: 10.1053/j.semnuclmed.2005.12.003. PMID 16517233
- [Background] Falk GL, Beattie J, Ing A, Falk SE, Magee M, Burton L, Van der Wall H. Scintigraphy in laryngopharyngeal and gastroesophageal reflux disease: a definitive diagnostic test? World J Gastroenterol. 2015 Mar 28;21(12):3619-27. doi: 10.3748/wjg.v21.i12.3619. PMID 25834329

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT05303298/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-20): https://cdn.clinicaltrials.gov/large-docs/98/NCT05303298/ICF_001.pdf